CLINICAL TRIAL: NCT05737537
Title: Blood Biomarkers Versus Blood Culture for Early Differentiation Between Fungal and Bacterial Infections in Pediatric Cancer Patients at South Egypt Cancer Institute
Brief Title: Using of Biomarkers and Blood Culture in Early Detection of Systemic Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mohammed Soliman Khalfallah, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: blood biomarkers in infections
Record Dates: First submitted 2023-01-23; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Invasive Fungal Infections
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infected pediatric cancer patients (Other)
  Interventions: Diagnostic Test: procalcitonin ,CRP and 1, 3- β -D- glucan in early diagnosis of invasive infections

INTERVENTIONS:
Diagnostic Test: procalcitonin ,CRP and 1, 3- β -D- glucan in early diagnosis of invasive infections — using of blood biomarkers (CRP ,procalcitonin and 1, 3- β -D- glucan) in early differentiation between fungal and bacterial infections in pediatric cancer patients in comparison to blood culture.

SUMMARY:
This work aims to:

1. Validate the performance of CRP, and PCT in early differentiating IFI from bacterial bloodstream infections.
2. Compare the results of CRP and PCT with the results of β-D- glucan. 3. Find the relationship between biomarkers levels [CRP, PCT and β-D- glucan] and the results of blood culture which is the gold standard of diagnosis.

DETAILED DESCRIPTION:
Immunocompromised children with cancer receiving chemotherapy or undergoing hematopoietic stem cell transplant (HSCT) are at high risk of infections. Invasive fungal infection (IFI) is a significant cause of morbidity and mortality. The incidence of IFI from 5.3% to 24% and the mortality rate from 18.6% to 67.6%. Definite diagnosis of fungal infection in immunocompromised patients is particularly challenging. However, the clinical presentation of IFI is not specific, especially in pediatric patients. The culture of blood is the major method to diagnose proven IFI, but the results are mostly negative, and culture is time consuming. New nonculture-based methods, including antigen-based assays, and molecular detection of fungal DNA which may allow early diagnosis and treatment of fungal infection. Molecular techniques, including DNA sequencing and polymerase chain reaction (PCR). These techniques have become more available in many laboratories; however, it lacks methodological standardization, and the results vary widely among laboratories. More attention paid to the biomarkers. 1, 3- β -D- glucan (BDG) is a component of the fungal cell wall and therefore it considered a pan-fungal detection method. Traditional biomarkers as C-reactive protein (CRP) and procalcitonin (PCT) have also been evaluated for their abilities in distinguishing IFI and other infections. In neonates, CRP levels were significantly higher in fungemia than in bacteremia, in adult patients, there was not a significant difference between the candidemia and bacteremia groups. The PCT value was markedly lower in the fungal infection group than in the bacteremia group at the onset of fever.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically suspected to have invasive fungal infections such as fever, cough or retrosternal pain, oral mucositis or perianal pain.
* Drug history of corticosteroids or chemotherapy.

Exclusion Criteria:

* Patients refuse to be part of the study.
* Patients have no symptoms of systemic infections.
* Drug history for antimicrobial before blood sample collection.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
comparison between levels of serum biomarkers (procalcitonin and CRP) and blood culture in differentiation between fungal and bacterial infections in immunocompromised children | early at the first 24 hours of symptoms of invasive infections
  study will be done on 90 participants. Blood samples will be collected under sterile conditions through a venipuncture.
  3-5 ml of blood will be collected on Bact alert bottles at the first 24 hours of fever early before taking antimicrobial treatment, cultured on blood agar. If positive, colonies will be cultured on McConkey, Mannitol salt agar and Sabouraud agar. Then the VITEK II method will be used to identify the colonies.
  At the same time 3 ml of blood will be incubated at room temperature for 30 minutes then centrifuged at 2500 rpm for 10 minutes then serum will be used for ELISA measurement of serum procalcitonin and β-D glucan.
  • Then trying to compare the results of blood culture with the biomarkers levels and find the relation between the results.

IPD SHARING:
Plan to Share IPD: Undecided